CLINICAL TRIAL: NCT00328133
Title: The Use of rFVIIa in Trauma Patients: A WTA/AAST Multi-Center Case Registry
Brief Title: The Use of rFVIIa in Trauma Patients: A Multi-Center Case Registry
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: Western Trauma Association (Other); Novo Nordisk A/S (Industry); American Association for the Surgery of Trauma (Other)
Responsible Party: Sponsor
Other Study IDs: H6693-27309-01
Record Dates: First submitted 2006-05-17; First posted 2006-05-19 (Estimated); Last update posted 2012-05-10 (Estimated); Status verified 2012-05

CONDITIONS: Traumatic Hemorrhage; Hemorrhagic Shock
Keywords: recombinant Factor VIIa; traumatic hemorrhage; hemorrhagic shock; coagulopathy
MeSH Terms: conditions — Shock, Hemorrhagic; Hemostatic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Trauma surgeons throughout the US have begun using recombinant activated factor VII (rFVIIa) to control severe hemorrhage following injury when traditional measures have failed. Despite promising results from several small studies, there remain several unanswered questions regarding the use of this relatively expensive product in injured patients including:

* The timing of administration
* Selection of appropriate patients who are most likely to benefit
* The effective dose in injured patients
* The potential need for repeated dosing
* The need for administration of platelets and correction of acidosis prior to administering the first dose
* The risks associated with the use of rFVIIa including venous and/or arterial thrombosis
* The potential for rFVIIa to cause or aggravate post-injury organ failure and/or infectious complications
* An analysis of cost versus benefit The purpose of this study is to collect a large sample of patients from multiple institutions in order to address the issues listed above. To this end, the Western Trauma Association Foundation is sponsoring a multi-center case registry for patients receiving rFVIIa for treatment of uncontrolled hemorrhage.

DETAILED DESCRIPTION:
This is a prospective, multi-center case registry that seeks to combine the collective experience with the use of rFVIIa at UCSF/SFGH with other trauma centers. The study is being conducted under the auspices of the Western Trauma Association and the American Association of the Surgery of Trauma. Both organizations have a long history of successfully completing multi-center studies. The outcomes to be used in this study are: 1) survival, 2) amount of blood products infused before and after rFVIIa, 3) coagulation factors (PTT, INR) before and after, and 4) the surgeon's assessment of hemostasis. Data will also be analyzed to determine the cost effectiveness of rFVIIa when compared with other methods of treating severe hemorrhage, primarily administration of blood products. Finally, the incidence of complications and thrombotic events after drug administration will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

Coagulopathy treated with rFVIIa

Exclusion Criteria:

none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective and prospective observational case review study on traumatically injured adult patients.
Sampling Method: Non-Probability Sample
Enrollment: 380 (Actual)
Dates: Start 2006-06; Primary Completion 2010-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Knudson, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco General Hospital, San Francisco, California, United States

REFERENCES:
- [Result] Knudson MM, Cohen MJ, Reidy R, Jaeger S, Bacchetti P, Jin C, Wade CE, Holcomb JB. Trauma, transfusions, and use of recombinant factor VIIa: A multicenter case registry report of 380 patients from the Western Trauma Association. J Am Coll Surg. 2011 Jan;212(1):87-95. doi: 10.1016/j.jamcollsurg.2010.08.020. Epub 2010 Nov 5. PMID 21115374